Title: Glutathione and Function in HIV patients

**NCT number: 02348775** 

Date submitted: February 2, 2021

## Statistical analysis plan

Baseline characteristics are summarized by means with standard deviations or frequencies with percentages. Controls were matched to PWH in a 1:1 ratio by age, sex, and BMI. A paired t-test was used to compare PWH and matched controls at baseline. A general linear mixed model was used to test for changes in outcomes across time points for PWH. The model included fixed effects for study time (discrete) and the matrix of correlated residuals assumed an unstructured format. The mixed model is used to estimate means with 95% confidence intervals and test the null hypothesis that there is no difference in means between time points. All hypothesis tests were assessed at the 0.05 level (two-sided). The p-values were not adjusted for multiple hypothesis testing due to the small sample size of this pilot study.